CLINICAL TRIAL: NCT05647044
Title: Neuromodulation for Impulsivity and Suicidality in Veterans With Mild Traumatic Brain Injury and Common Co-occurring Mental Health Conditions
Brief Title: Frontal iTBS for Impulsivity and Suicidal Ideation in Veterans With Mild Traumatic Brain Injury
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4298-W
Record Dates: First submitted 2022-11-15; First posted 2022-12-12 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Mild Traumatic Brain Injury; Suicidal Ideation; Impulsivity
Keywords: brain concussion; brain injuries, traumatic; brain injuries; self-injurious behavior; suicide, attempted; suicide; impulsive behavior; risk-taking; brain diseases; craniocerebral trauma; social problems; mental disorders
MeSH Terms: conditions — Brain Concussion; Suicidal Ideation; Impulsive Behavior; Brain Injuries, Traumatic; Brain Injuries; Self-Injurious Behavior; Suicide, Attempted; Suicide; Risk-Taking; Brain Diseases; Craniocerebral Trauma; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Magventure MagProX100 with MagOption stimulator and Magpro Cool Coil B65 A/P and Magpro C-B60
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be a triple blinded study with participants, investigators and outcomes assessors all masked until study completion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- active iTBS (Active Comparator): Subjects receiving active iTBS treatment
  Interventions: Device: intermittent theta burst stimulation
- placebo iTBS (Placebo Comparator): Subjects receiving placebo (sham) iTBS treatment
  Interventions: Device: placebo intermittent theta burst stimulation

INTERVENTIONS:
Device: intermittent theta burst stimulation — intermittent theta burst stimulation (iTBS) will be delivered with the Magventure MagProX100 with MagOption stimulation and Magpro Cool Coil B65 A/P. The Magpro Cool Coil B65 A/P can be switched to active or placebo. The Magventure C-B60 coil will be used to deliver single TMS pulses for motor threshold determination.
  Other Names: iTBS
  Arms: active iTBS
Device: placebo intermittent theta burst stimulation — intermittent theta burst stimulation (iTBS) will be delivered with the Magventure MagProX100 with MagOption stimulation and Magpro Cool Coil B65 A/P. The Magpro Cool Coil B65 A/P can be switched to active or placebo. The Magventure C-B60 coil will be used to deliver single TMS pulses for motor threshold determination.
  Other Names: placebo iTBS
  Arms: placebo iTBS

SUMMARY:
The investigators hope to develop a treatment for suicidal ideation (SI), impulsivity and functional impairments (such as difficulties in social and work settings) that occur after a mild traumatic brain injury (mTBI). These conditions have been shown to be linked. The investigators are using a high-powered magnetic pulse, called intermittent theta burst stimulation (iTBS) applied to the head to see if it can improve these symptoms. The high-powered magnetic pulse causes certain cells in the brain to activate, which seems to strengthen connections between parts of the brain. The purpose of this research is to gather early information on the safety and effectiveness of iTBS provided to the front of the head for impulsivity, SI and functional deficits after mTBI. The investigators plan to use the data collected in this study to develop larger studies in the future. iTBS is FDA approved, but not for these specific symptoms, or in the specific location the investigators are placing it. The investigators are testing to see if its effective for the above conditions when applied to the front of the head.

DETAILED DESCRIPTION:
Individuals with mild traumatic brain injury (mTBI) are at increased risk of dying by suicide compared to those without - both among Veteran and civilian populations. 22% of Veterans with mTBI report struggling with suicidal ideation (SI). Despite this, there are no effective evidence-based treatments for co-occurring mTBI and SI. Deficits in social and occupational functioning, which often follow mTBI, are strongly related to suicidal ideation (SI) and improvements in these areas are known to lessen SI. Thus, improving function for those with mTBI and SI is of great potential significance. The impulsivity that Veterans with mTBI exhibit is referred to as "negative urgency impulsivity". It often involves aggressive and self-harming behaviors, which impede societal re-integration and rehabilitation. Prior studies indicate negative urgency impulsivity is: (1) a common TBI sequela and (2) a risk factor for SI. Previous studies have also indicated individuals with TBI, SI and negative urgency impulsivity had reduced right-sided ventromedial prefrontal cortex (VMPFC) volume compared to Veterans without these conditions. The VMPFC plays a key role in controlling impulsive limbic responses. These findings are consistent with published reports suggesting individuals with reduced VMPFC volume are more likely to (a) have SI and (b) behave impulsively.

Transcranial magnetic stimulation (TMS) holds significant therapeutic promise for post-mTBI SI, impulsivity and functional deficits. TMS induces neuroplasticity, leading to changes that have the potential to improve neurorehabilitation outcomes. TMS is effective for treating post-TBI depression when administered to the dorsolateral prefrontal cortex. Intermittent theta burst stimulation (iTBS) is a "second generation" form of TMS that is delivered more rapidly. It has been proposed that frontal pole TMS could directly strengthen connections throughout the prefrontal cortex, including the VMPFC, thereby dampening limbic system activity. Such a TMS treatment strategy could be used to treat post-mTBI impulsivity and SI, ultimately allowing Veterans to regain functioning. It is not know which Veterans would benefit most from this treatment; examining neural connectivity changes before and after iTBS could determine who would respond to frontal pole iTBS and why.

The investigators will conduct a randomized, double-blinded frontal iTBS pilot clinical trial for Veterans with mTBI, impulsivity and SI. As this is a novel treatment approach for this population, this project will focus on testing the safety, feasibility and tolerability of frontal pole iTBS. To inform future research, this project will determine the preliminary effects of iTBS on functioning, negative urgency impulsivity and SI among the pilot sample. This project will also inform future research by examining the relationships between the functional neural connectivity of the VMPFC to the limbic system and how this is affected by iTBS using resting state functional connectivity (rsFC) neuroimaging data, pre- and post-iTBS.

ELIGIBILITY:
Inclusion Criteria:

* 22-65 years of age
* can read and speak English
* meets criteria for mTBI according to the symptom attribution and classification (SACA) scale
* Has a C-SSRS (suicidal ideation rating) of >1 within the past month
* Has a history of impulsivity documented in the medical chart and/or a score of >20 on the UPPS-P negative urgency impulsivity subscale

Exclusion Criteria:

* Has contraindications to iTBS (i.e., epilepsy)
* Has contraindications to MRI (i.e., claustrophobia, ferromagnetic metal implants)
* Has an active substance use disorder per the DSM-V criteria
* Has a history of moderate to severe TBI
* Has a history of non-traumatic neuroinjury (i.e., stroke, neurosurgery, hemorrhage)
* Has a history of, or current psychosis not due to an external cause
* Is pregnant
* Has an active, unstable medical condition
* Is within 12 weeks of a major surgery or operation
* Is within 1 year of TBI

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Session Completion Rate | Endpoint - after last iTBS session, approximately 2 weeks
  For establish intervention feasibility and tolerability, the study will tract the number of completed iTBS sessions and compute completion percentage rates for each participant.
Change in Social and Occupational Functioning Assessment Scale (SOFAS) | Rated at baseline, study midpoint (at the end of week 1) and study completion, approximately 2 weeks after study begins
  The Social and Occupational Functioning Assessment scale is a rating, given by a trained medical provider, of an individual's ability to perform basic functioning (such as hygiene, maintaining a job, having social relationships). The scale is from 10, meaning unable to function without harming self or others, to 100, meaning superior functioning in all areas. The investigators will be assessing this at subject's baseline, after 1 week of treatment (5 treatment sessions, at the end of week 1) and at study completion (approximately 2 weeks after study starts) to see if there is a change over time in this measure.

SECONDARY OUTCOMES:
Change in Columbia Suicide severity rating scale (C-SSRS) | Rated at baseline, study midpoint (at the end of week 1) and study completion, approximately 2 weeks after study begins.
  The C-SSRS is a short questionnaire addressing any recent suicidal thoughts or behaviors that have occurred. A score of 0 means there have been no suicidal thoughts or behaviors, anything above a 0 means some element of suicidality has been experienced by the test-taker. The investigators will be assessing this at subject's baseline, after 1 week of treatment (5 treatment sessions, at the end of week 1), and at study completion (approximately 2 weeks after study starts) to see if there is a change over time in this measure.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra L Aaronson, MD, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified data set will be created and shared. Final data sets will be made available as per Hines VA Hospital local policy for long term storage and access until enterprise-level resources become available. These data will be available upon request by researchers and scientists in accordance with federal guidelines and Hines local policy.
  The data provided will be sufficient for anyone to perform analogous or supplemental analyses that would permit validation of the analysis and results. The sharing of data will enable others to evaluate the data and to validate and interpret the data independently. In order to ensure that replication is possible and transparency, statistical code complementary to datasets will be made available through the Federal Interagency Traumatic Brain Injury Research Informatics System
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: After primary publication of study data
Access Criteria: The data will be available upon request by researchers and scientists in accordance with federal guidelines and local policy.
URL: https://fitbir.nih.gov/

REFERENCES:
- [Derived] Bernanke A, Hasley R, Sabetfakhri N, de Wit H, Smith BM, Wang L, Brenner LA, Hanlon C, Philip NS, Ajilore O, Herrold A, Aaronson A. Frontal Pole Neuromodulation for Impulsivity and Suicidality in Veterans With Mild Traumatic Brain Injury and Common Co-Occurring Mental Health Conditions: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2024 Dec 13;13:e58206. doi: 10.2196/58206. PMID 39671573